CLINICAL TRIAL: NCT03486327
Title: Transabdominal Ultrasound With BR55 for Characterization of Pancreatic Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision; expiration of available study agent due to long recruitment timeline.
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: BR55-110
Record Dates: First submitted 2018-03-02; First posted 2018-04-03 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Up to 24 subjects will be enrolled into 3 dose groups starting with the lowest dose group as follows: Dose group 0.03mL/kg, dose group 0.05mL/kg and dose group 0.08mL/kg/, with a maximum of 8 patients in each dose group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.03mL/kg Dose Group (Experimental): A group of up to 8 subjects to receive a single dose of BR55 at 0.03mL/kg.
  Interventions: Drug: BR55
- 0.05mL/kg Dose Group (Experimental): A group of up to 8 subjects to receive a single dose of BR55 at 0.05mL/kg.
  Interventions: Drug: BR55
- 0.08mL/kg Dose Group (Experimental): A group of 8 subjects to receive a single dose of BR55 at 0.08mL/kg.
  Interventions: Drug: BR55

INTERVENTIONS:
Drug: BR55 — A novel targeted ultrasound contrast agent

SUMMARY:
This is an exploratory, single center, open label, parallel-dose, and prospective study of BR55 contrast-enhanced ultrasonography (CEUS) for characterization of solid pancreatic lesions in subjects with suspected pancreatic ductal adenocarcinoma (PDAC) using transabdominal US.

DETAILED DESCRIPTION:
Approximately twenty-four (24) subjects with suspected PDAC and scheduled to undergo surgical resection within 30 days (but not before 24 hours) after the transabdominal BR55 CEUS examination will be enrolled into 3 dose groups, 0.03, 0.05, and 0.08 mL/kg, with a maximum of 8 patients in each dose group.

ELIGIBILITY:
Inclusion Criteria:

Enroll a subject in this study if the subject meets the following inclusion criteria:

* Is at least 18 years of age;
* Has at least one solid pancreatic lesion;
* Is scheduled to undergo surgical resection for suspected PDAC not earlier than 24 hours and not later than 30 days following BR55 administration;
* Provides written Informed Consent and is willing to comply with protocol requirements.

Exclusion Criteria:

Exclude a subject from this study if the subject does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Is a pregnant or lactating female. Exclude the possibility of pregnancy:

  * by testing on site at the institution (serum βHCG) within 24 hours prior to the start of investigational product (IP) administration,
  * by surgical history (e.g., tubal ligation or hysterectomy),
  * by post-menopausal status with a minimum 1 year without menses;
* Has undergone prior systemic therapy for pancreatic cancer;
* Has history of any concurrent malignancy;
* Has history of any clinically unstable cardiac condition including class III/IV congestive heart failure;
* Has had any severe cardiac rhythm disorders within 7 days prior to enrolment;
* Has severe pulmonary hypertension (pulmonary artery pressure > 90mmHg) or uncontrolled systemic hypertension and/or respiratory distress syndrome;
* Has open and/or non-healing wounds in the chest, abdomen and pelvis;
* Has other systemic vascular abnormalities associated with neovascularization, such as macular degeneration, that in the opinion of the investigator could significantly affect the ability to evaluate the effects of BR55;
* Is participating in a clinical trial or has participated in another trial with an investigational compound within the past 30 days prior to enrolment;
* Has previously been enrolled in and completed this study;
* Has any known allergy to one or more of the ingredients of the IP or to any other contrast media;
* Is determined by the Investigator that the subject is clinically unsuitable for the study;
* Has had major surgery, including laparoscopic surgery within 3 months prior to enrolment;
* Has history of pancreatic surgery (e.g., cyst removal);
* Has acute pancreatic abnormalities (acute pancreatitis or trauma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As of July 31, 2021, enrollment was terminated for Study BR55-110 due to expiration of available BR55. Therefore, only 4 participants were enrolled in the first cohort of this study (0.03 mL/kg). No participant was enrolled in the 0.05 mL/kg or 0.08 mL/kg groups.
Groups:
- 0.05mL/kg Dose Group: A group of up to 8 subjects to receive a single dose of BR55 at 0.05mL/kg.
  BR55: A novel targeted ultrasound contrast agent
  No study participant was enrolled in this group.
- 0.08mL/kg Dose Group: A group of 8 subjects to receive a single dose of BR55 at 0.08mL/kg.
  BR55: A novel targeted ultrasound contrast agent
  No study participant was enrolled in this group.
Period: Overall Study
Arm/Group | 0.03mL/kg Dose Group | 0.05mL/kg Dose Group | 0.08mL/kg Dose Group
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As of July 31, 2021, enrollment was terminated for Study BR55-110 due to expiration of available BR55. Therefore, only 4 participants were enrolled in the first cohort of this study (0.03 mL/kg). No participant was enrolled in the 0.05 mL/kg or 0.08 mL/kg groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.03mL/kg Dose Group | 0.05mL/kg Dose Group | 0.08mL/kg Dose Group | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 1 |  |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [60 to 78] |  |  | 65.5 [60 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 4 |  |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  |  | 1
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  |  | 4
Total Volume (mL) Injected [Mean (Full Range); unit: mL] | 2.00 [1.60 to 2.37] |  |  | 2.00 [1.60 to 2.37]

OUTCOME MEASURES:

1. Primary Outcome: 1. Visual Assessment of Enhancement
Description: BR55-enhanced images will be visually assessed using a 3-point scale (no enhancement, weak enhancement, strong enhancement).
Time Frame: Up to 24 hours post-dose on Day 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 0.03mL/kg Dose Group | 0.05mL/kg Dose Group | 0.08mL/kg Dose Group
Number analyzed (Participants) | 4 | 0 | 0
Participants
  No enhancement | 0 |  |
  Weak enhancement | 3 |  |
  Strong enhancement | 1 |  |

2. Primary Outcome: 2. Adverse Events
Description: Number of participants who received the contrast agent and experienced an adverse event.
Time Frame: From the time of signing Informed Consent through 24 hours post-dose, up to a maximum of 11 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 0.03mL/kg Dose Group | 0.05mL/kg Dose Group | 0.08mL/kg Dose Group
Number analyzed (Participants) | 4 | 0 | 0
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety monitoring began at the time of signing Informed Consent and continued for 24 hours after BR55 administration, up to a maximum of 11 days.
Description: As of July 31, 2021, enrollment was terminated for Study BR55-110 due to expiration of available BR55. Therefore, only 4 participants were enrolled in the first cohort of this study (0.03 mL/kg). No participant was enrolled in the 0.05 mL/kg or 0.08 mL/kg groups.
Arm/Group | 0.03mL/kg Dose Group | 0.05mL/kg Dose Group | 0.08mL/kg Dose Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03mL/kg Dose Group (N=4) | 0.05mL/kg Dose Group (N=0) | 0.08mL/kg Dose Group (N=0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Cheek L pruritus
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03486327/Prot_SAP_000.pdf